CLINICAL TRIAL: NCT01180946
Title: Vitamin D Deficiency in Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sherri-Ann M. Burnett-Bowie, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2010-P-001126/1
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Healthy; Vitamin D Deficiency
Keywords: FGF23; FGF-23; vitamin D; vitamin D deficiency; insulin resistance; Healthy volunteers
MeSH Terms: conditions — Vitamin D Deficiency; Insulin Resistance | interventions — Ergocalciferols; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ergocalciferol (Active Comparator): Weekly ergocalciferol for 16 weeks
  Interventions: Dietary Supplement: ergocalciferol
- Placebo (Placebo Comparator): Placebo pill. Note that all subjects in this arm will receive vitamin D repletion at the conclusion of the study.
  Interventions: Other: placebo pill

INTERVENTIONS:
Dietary Supplement: ergocalciferol — ergocalciferol (a dietary form of vitamin D). 50,000 units by mouth once a week for 16 weeks.
  Other Names: vitamin D
  Arms: Ergocalciferol
Other: placebo pill — placebo pill once weekly for 16 weeks. At the end of the study, subjects in this arm will receive vitamin D repletion
  Arms: Placebo

SUMMARY:
Fibroblast growth factor 23 (FGF23) is a newly discovered hormone which regulates phosphate and vitamin D levels. In this study, we are looking at what the normal levels of FGF23 are in adolescent girls and how these levels vary with other hormonal measurements. We will also be looking at whether vitamin D supplementation in adolescents who are deficient in vitamin D alters the levels of FGF23 and other factors including insulin resistance.

DETAILED DESCRIPTION:
Fibroblast growth factor 23 (FGF23) is a newly discovered hormone. Its primary function is to regulate phosphate metabolism, which it does both by directly regulating phosphate excretion through the kidney as well as by regulating vitamin D activity. What controls FGF23 levels is still under investigation; potential factors include dietary phosphate intake and vitamin D levels.

In this pilot study, we aim to investigate what the normal levels of FGF23 are in healthy girls and how these are related to other measurements of bone and mineral metabolism. Since vitamin D deficiency is very common in healthy girls, we expect a subset of the subjects in this study to be vitamin D deficient. We will then randomize these girls to vitamin D repletion or placebo and follow changes in FGF23 levels. Vitamin D deficiency has also been implicated in insulin resistance which is a precursor to diabetes. We will therefore also look at changes in insulin resistance with vitamin D repletion.

ELIGIBILITY:
Inclusion Criteria:

* healthy girls aged 9-18 years

Exclusion Criteria:

* significant cardiac, hepatic, oncologic, or psychiatric disease
* a history of malabsorption, kidney stones, hypoparathyroidism, or growth hormone deficiency
* pregnancy
* diabetes mellitus
* BMI>/= 99th percentile for age and sex
* fracture within the preceding 3 months
* hypogonadism (no pubertal development by age 12, absence of menarche by age 14)
* serum calcium <8 mg/dl or >11 mg/dl
* radiographic evidence of rickets
* use of medications know to affect serum phosphate levels including phosphate-binding antacids, sodium etidronate, calcitonin, excessive doses of vitamin D (>1000 units per day), excessive doses of vitamin D (>20,000 units/day), calcitriol, growth hormone, or anti-convulsants.
* use of hormonal birth control

Ages: 9 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2010-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
change in FGF23 level with vitamin D repletion | baseline and 16 weeks

SECONDARY OUTCOMES:
change in bone turnover markers with vitamin D repletion | baseline and 16 weeks
change in mineral metabolism factors with vitamin D repletion | baseline and 16 weeks
change in insulin sensitivity with vitamin D repletion | baseline and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sherri-Ann Burnett-Bowie, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Burnett-Bowie SM, Henao MP, Dere ME, Lee H, Leder BZ. Effects of hPTH(1-34) infusion on circulating serum phosphate, 1,25-dihydroxyvitamin D, and FGF23 levels in healthy men. J Bone Miner Res. 2009 Oct;24(10):1681-5. doi: 10.1359/jbmr.090406. PMID 19419295
- [Background] Burnett-Bowie SM, Mendoza N, Leder BZ. Effects of gonadal steroid withdrawal on serum phosphate and FGF-23 levels in men. Bone. 2007 Apr;40(4):913-8. doi: 10.1016/j.bone.2006.10.016. Epub 2006 Dec 8. PMID 17157573
- [Background] Burnett SM, Gunawardene SC, Bringhurst FR, Juppner H, Lee H, Finkelstein JS. Regulation of C-terminal and intact FGF-23 by dietary phosphate in men and women. J Bone Miner Res. 2006 Aug;21(8):1187-96. doi: 10.1359/jbmr.060507. PMID 16869716
- [Derived] Mitchell DM, Juppner H, Burnett-Bowie SM. FGF23 Is Not Associated With Age-Related Changes in Phosphate, but Enhances Renal Calcium Reabsorption in Girls. J Clin Endocrinol Metab. 2017 Apr 1;102(4):1151-1160. doi: 10.1210/jc.2016-4038. PMID 28323960